CLINICAL TRIAL: NCT05501691
Title: Effect of Low-Level Diode Laser on Dentin Topography And Sensitive Non-Carious Cervical Lesions Prior to Composite Restoration, And Dentin Bonding And Clinical Durability of Composite Restorations (A Two Year Split-mouth Randomized Controlled Trial)
Brief Title: Effect of Diode Laser on Sensitive NCCLs Prior to Composite Restoration, Dentin Bonding, and Clinical Durability of Composite Restorations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Raghda Hegazy, Principal Investigator, Alexandria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0048-06/2022; IORG0008839 (Other: International No: Alexandria University)
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: In this randomized controlled clinical trial, patients with NCCLs will be included (four teeth in each participant). The teeth will be randomly assigned into four groups according to diode laser irradiation wavelength Group 1 (placebo) laser simulation, Group 2 (445 nm) diode laser wavelength, Group 3 (660 nm) diode laser wavelength, and Group 4 (970 nm) diode laser wavelength.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The allocation will be hidden from patients, and they will not know which teeth are lased and which will receive the placebo treatment. In addition, for blinding, the restoration procedure is performed by one person, and the cold test is performed by another person who is unaware of the distribution. Furthermore, the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Laser Simulation
  Interventions: Other: Placebo
- 445 nm (Experimental): 445 nm Diode Laser Wavelength (SiroLaser Blue)
  Interventions: Radiation: 445 nm Diode Laser Wavelength
- 660 nm (Experimental): 660 nm Diode Laser Wavelength (SiroLaser Blue)
  Interventions: Radiation: 660 nm Diode Laser Wavelength
- 970 nm (Experimental): 970 nm Diode Laser Wavelength (SiroLaser Blue)
  Interventions: Radiation: 970 nm Diode Laser Wavelength

INTERVENTIONS:
Other: Placebo — Laser Simulation
  Arms: Placebo
Radiation: 445 nm Diode Laser Wavelength — Irradiated Using a 445 nm Diode Laser Wavelength
  Arms: 445 nm
Radiation: 660 nm Diode Laser Wavelength — Irradiated Using a 660 nm Diode Laser Wavelength
  Arms: 660 nm
Radiation: 970 nm Diode Laser Wavelength — Irradiated Using a 970 nm Diode Laser Wavelength
  Arms: 970 nm

SUMMARY:
This study will investigate the efficacy of three diode laser wavelengths 445 nm, 660 nm, 970 nm when applied just before placement of composite restoration on reducing postoperative sensitivity from Non-carious cervical lesions (NCCLs) with class V cavity preparation.

DETAILED DESCRIPTION:
In this randomized clinical trial, patients with NCCLs will be included (four teeth in each participant). After class V cavity preparation in the NCCLs, the teeth will be randomly assigned into four groups according to diode laser irradiation wavelength Group 1 (placebo) laser simulation and Group 2 (445 nm) diode laser wavelength, Group 3 (660 nm) diode laser wavelength, and Group 4 (970 nm) diode laser wavelength. Following laser irradiation, the universal self-etch adhesive will be applied and all the cavities will be restored with the same resin composite. Tooth sensitivity to a cold stimulus will be recorded using a visual analogue scale (VAS) before treatment and on follow-up days 1, 14 followed by 1, 3, and 6 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. NCCLs on the Buccal Surface of Teeth, Maxilla, or Mandible.
2. Preoperative VAS Score > 2.
3. Good Oral Hygiene. Score (0-1.2).
4. Teeth Must be Vital.

Exclusion Criteria:

1. Teeth with a History of Trauma, Dental caries, Defective Restoration, Pulpitis, Occlusal Restoration.
2. Teeth with Periodontal Disease or History of Surgical Procedure.
3. Use of Desensitizing Toothpaste or Solutions in the Past 3 Month.
4. Patients Taking Analgesics within 72 h Before Sensitivity Testing.
5. Patients with Known Allergic Reactions Against Any Material to be Used.
6. Patients with a History of Psychological Diseases and those Taking Antipsychotic Medications.
7. Pregnancy or Nursing.
8. Unwillingness of the Patient to the Treatment Procedure.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Dentin Hypersensitivity Assessed from Baseline to After Exposure to Diode Laser Radiation. | Change in Pain Scores From Baseline on the Visual Analog Scale at Day 1, Day 14, Followed by 1,3, and 6 Month Postoperatively.
  Dentin Hypersensitivity is Determined using Cold Stimulus. Utilizing Visual Analog Scale (VAS) Reading 0-10 Where 0 is No Pain, While 10 is the Most Experienced Pain.

SECONDARY OUTCOMES:
Clinical assessment for esthetic, functional, and biological responses to restorative materials. | Time frame: Restorations are evaluated for esthetic, functional, and biological properties over follow-up periods of 6 months, 12 months, and 24 months.
  The restoration's esthetic assessment includes 1. surface luster, 2. surface staining, and 3. color stability and translucency.
  The functional assessment of the restoration includes 1. fracture and retention, 2. marginal adaptation, 3. wear, and 4. the patient's view
  . The biological category, ratings include 1. Postoperative sensitivity or hypersensitivity and tooth vitality, 2. Recurrence of carious, erosion, abrasion 3. Tooth integrity (enamel cracks) 4. Periodontal response 5. Adjacent mucosa 6. Oral and general health.
  Each criterion will be scored 1-5. Each score represents 1. clinically excellent/ very good, 2. clinically good, 3. clinically sufficient/ satisfactory, 4. clinically unsatisfactory, and 5. clinically poor.

CONTACTS AND LOCATIONS:
Overall Officials: Raghda A Hegazy, Bachelor, Principal Investigator — Pharos University; El Sayed M Mahmoud, Professor, Study Chair — Alexandria University; Ahmed A Holiel, Lecturer, Study Director — Alexandria University
Locations (1):
- Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hegazy RA, Mahmoud EM, Holiel AA. EFFECT OF LOW-LEVEL DIODE LASER ON DENTIN TOPOGRAPHY AND SYMPTOMATIC NONCARIOUS CERVICAL LESIONS PRIOR TO COMPOSITE RESTORATIONS: A SPLIT-MOUTH RANDOMIZED CONTROLLED TRIAL. J Evid Based Dent Pract. 2024 Jun;24(2):101969. doi: 10.1016/j.jebdp.2024.101969. Epub 2024 Jan 17. PMID 38821658